CLINICAL TRIAL: NCT06615375
Title: Phase 2b, Double-blind, Placebo-controlled Efficacy Challenge Study With the Shigella Tetravalent Bioconjugate Vaccine Shigella4V2
Brief Title: A Human Challenge Study to Assess Protection of a Shigella Tetravalent Bioconjugate Vaccine
Acronym: S4V03
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LimmaTech Biologics AG (Industry)
Collaborators: Emory University (Other); Johns Hopkins Bloomberg School of Public Health (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S4V03
Record Dates: First submitted 2024-09-20; First posted 2024-09-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Shigellosis
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Shigella4V2 High dose (Experimental): 1 injection of high dose Shigella4V2 and 1 injection of low dose Shigella4V2 will be injected intramuscularly in the deltoid muscle
  Interventions: Biological: Shigella4V2
- Shigella4V2 Low dose (Experimental): 2 injections of low dose of Shigella4V2 will be injected intramuscularly in the deltoid muscle
  Interventions: Biological: Shigella4V2
- Placebo (Placebo Comparator): 2 injections of PBS will be injected intramuscularly in the deltoid muscle
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Shigella4V2 — Shigella4V2 is a tetravalent bioconjugate vaccine
  Arms: Shigella4V2 High dose; Shigella4V2 Low dose
Biological: Placebo — Phosphate-buffered saline
  Arms: Placebo

SUMMARY:
In this challenge study, the bioconjugate candidate vaccine Shigella4V2 will be tested for its ability to induce an immune response that protects healthy adult volunteers from infection with a wild-type Shigella sonnei strain compared to participants receiving placebo.

DETAILED DESCRIPTION:
The tetravalent Shigella4V2 bioconjugate vaccine candidate will be tested for safety and preliminary efficacy in a Phase 2b controlled human infection model (CHIM) study at three sites in the United States. This trial will be conducted as a parallel-group, randomized, double-blind, multicenter, placebo-controlled study to evaluate the safety, immunogenicity, and efficacy of two injections of Shigella4V2 in healthy Shigella naïve participants 18-50 years of age, with the second injection administered one month before challenge with S. sonnei 53G strain. It will have two steps:

1. Step 1, a dose confirmation step, in which a first injection of Shigella4V2 (high dose or low dose, adjuvanted with Alhydrogel) will be administered alongside a placebo arm (phosphate-buffered saline) at a ratio of 2:2:1. A second injection of either Shigella4V2 low dose or placebo will be administered about 6 months after the first injection.
2. Step 2, in which participants will be randomized to the Shigella4V2 dose selected after Step 1 or to placebo at a ratio of 1:1. Participants will receive two injections, 28 days apart. One month after the second injection, they will be challenged with 1500 CFU of the virulent Shigella sonnei strain 53G.

ELIGIBILITY:
Inclusion Criteria:

Step 1 and Step 2:

1. Age 18-50 years (inclusive).
2. In good health and stable medical condition, determined by MH, laboratory results, and physical examination during screening period.
3. Negative pregnancy test at the time of 1st injection, for participants of childbearing potential.
4. Persons of childbearing potential must agree to avoid pregnancy by use of effective contraception for 30 days prior to 1st injection and throughout the study. Participants assigned female at birth and unable to bear children must have this documented (e.g., tubal ligation or hysterectomy).
5. Willingness to participate in the study after all aspects of the protocol have been explained and written informed consent obtained.
6. Availability for the study duration, including all planned follow-up visits and phone calls.
7. Willingness to refrain from participating in other studies of investigational products until completion of the last study contact.

   Step 2 only:
8. Demonstrated comprehension of the protocol procedures, knowledge of Shigella- associated illness, and passing score of 70% or better on a comprehension assessment. Maximum two attempts are allowed.

Exclusion Criteria:

Step 1 and Step 2:

1. Participants currently pregnant, lactating, or intending to become pregnant during the study period as reported by the participant.
2. Presence of a significant medical or psychiatric condition which in the opinion of the investigator precludes participation in the study.
3. Clinically significant abnormalities in vital signs or in screening hematology / blood chemistry as determined by the investigator.
4. Presence in the serum of HIV 1/2 antibody, HBs-Ag, or HCV antibody (if confirmed positive by Hepatitis C confirmatory test, i.e., recombinant immunoblot assay (RIBA), polymerase chain reaction (PCR)).
5. Evidence of current excessive alcohol consumption or drug dependence (e.g. according to medical history).
6. Known or suspected impairment of immunological function (e.g., documented HIV infection, asplenia/splenectomy, or history of autoimmune disease or lymphoproliferative disorder).
7. BMI < 19 or > 35 kg/m2.
8. Recent vaccination or planned vaccination within 14 days of 1st study injection for inactivated vaccines and within 30 days for live vaccines.
9. Recent receipt of an investigational product within 30 days preceding the 1st study injection or planned during the entire study period.
10. Recent treatment with immunoglobulins or blood products within 3 months preceding the 1st study injection or planned use during the entire study period.
11. Use of any medication known to affect the immune function (e.g., systemic steroids) within 30 days preceding the 1st study injection or planned use during the entire study period.
12. Symptoms consistent with Traveler's Diarrhea concurrent with travel to countries where Shigella infection is endemic (most of the developing world).
13. Vaccination for or ingestion of Shigella.
14. Use of systemic antibiotics during the 7 days before 1st injection.
15. Serum IgG titers to S. sonnei LPS ≥ 2500.
16. Current occupation involving the handling of Shigella bacteria.
17. History of allergy to components of the study vaccine (Alhydrogel), to placebo (PBS), or to soy, or any other allergy the investigator deems to increase their risk of AEs in the study.
18. Any other criteria which, in the investigator's opinion, would compromise the ability of the participant to participate in the study, the safety of the study, or the results of the study.
19. Part of study personnel or close family member of personnel conducting the study.

    Step 2 only:
20. Personal history of inflammatory ReA.
21. Positive blood test for HLA-B27 antigen.
22. Personal history of IBS as defined by Rome IV criteria.
23. Regularly abnormal stool pattern (fewer than 3 per week or more than 3 per day).
24. Regular use of laxatives, antacids, or other agents to lower stomach acidity.
25. Known allergy to challenge agent components.
26. Known allergy to ciprofloxacin or trimethoprim-sulfamethoxazole.
27. Evidence of IgA deficiency (serum IgA < 7 mg/dL or limit of detection of assay).
28. Planning to travel to Shigella endemic countries before completion of the challenge phase of the study.
29. Personal history of inflammatory bowel disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that the Shigella4V2 bioconjugate vaccine protects against shigellosis following challenge with the wild type S. sonnei 53G strain. | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccinees vs. placebo
  The number of challenged participants with shigellosis post-challenge during the inpatient period that received vaccine compared to participants who received placebo. Shigellosis is defined as:
  1. Severe diarrhea; OR
  2. Moderate diarrhea AND [fever OR ≥ 1 at least moderate constitutional/enteric symptoms OR ≥ 2 episodes of vomiting in 24 h]; OR
  3. Dysentery AND [fever OR ≥ 1 at least moderate constitutional/enteric symptoms OR ≥ 2 episodes of vomiting in 24 h]

SECONDARY OUTCOMES:
The number of challenged participants with shigellosis post-challenge during the inpatient period that responded to Shigella4V2 vaccine compared to participants who received placebo. | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo
  Occurrence of shigellosis among the challenged participants that responded from the time of challenge until the end of the inpatient monitoring period
Efficacy - Number of participants with moderate-to-severe shigellosis | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Occurrence of moderate-to-severe shigellosis post-challenge during the inpatient period. Moderate-to-severe shigellosis is defined as:
  1. Moderate or severe diarrhea AND [fever OR ≥ 1 severe constitutional/enteric symptoms OR ≥ 3 episodes of vomiting in 24 h]; OR
  2. Dysentery AND [fever OR ≥ 1 severe constitutional/enteric symptoms OR ≥ 3 episodes of vomiting in 24 h]
Efficacy - Number of participants with diarrhea of any severity | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Occurrence of ≥ 2 loose stools in any 24-hour period post-challenge during the inpatient period
Efficacy - Number of participants with severe diarrhea | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Occurrence of ≥ 6 loose stools or more than 800 g of stool in any 24-hour period post-challenge during the inpatient period
Efficacy - Number of participants with moderate or severe diarrhea | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Occurrence of ≥ 4 loose stools or ≥ 400 g of stool in any 24-hour period post-challenge during the inpatient period
Efficacy - Number of participants with more severe diarrhea | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Occurrence of ≥ 10 loose stools or ≥ 1000 g of stool in any 24-hour period post-challenge during the inpatient period
Efficacy - Maximum weight of grade 3-5 stools passed in 24 h per participant | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Maximum weight of loose stools (grade 3-5) passed in any 24-hour period post-challenge during the inpatient period
Efficacy - Maximum number of grade 3-5 stools passed in 24 h per participant | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Maximum number of loose stools (grade 3-5) passed in any 24-hour period post-challenge during the inpatient period
Efficacy - Number of participants with moderate or severe constitutional enteric symptoms | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Occurrence of moderate or severe constitutional enteric symptoms post-challenge during the inpatient period
Efficacy - Number of participants with severe constitutional enteric symptoms | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Occurrence of severe constitutional enteric symptoms post-challenge during the inpatient period
Efficacy - Number of participants with fever | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Occurrence of fever post-challenge during the inpatient period
Efficacy - Highest recorded temperature | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Highest recorded temperature post-challenge during the inpatient period
Efficacy - Time from challenge to onset of diarrhea | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Time (in hours) from challenge to first loose stool that contributes to diarrhea (≥ 2 loose stools in a 24-hour period)
Efficacy - Time from challenge to onset of shigellosis | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Time (in hours) from challenge to first event (e.g., first loose stool, first day of fever or moderate symptom, or first episode of vomiting) that contributes to the shigellosis endpoint
Efficacy - Duration of diarrhea | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Duration will be calculated as the time (in hours) from the first stool that contributes to diarrhea until the last stool that contributes to diarrhea, occurring post-challenge during the inpatient period, irrespective of intermittent time without loose stools
Efficacy - Shigella disease severity score | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Shigella disease severity score (scale from 0 to 9) post-challenge during the inpatient period
Efficacy - Number of participants requiring early antibiotic therapy | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Receipt of antibiotic therapy prior to 5 days after challenge
Efficacy - Number of participants requiring IV fluids | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccine responders vs. placebo as well as vaccinees vs. placebo
  Receipt of IV fluids post-challenge during the inpatient period
Efficacy - Number of participants with blood in stool as confirmed by hemoccult | To be evaluated post-challenge during the inpatient period (Day 56 through Day 65) in vaccinees vs. placebo
  Occurrence of at least one stool with blood as confirmed by hemoccult post-challenge during the inpatient period
Safety - Solicited Local and Systemic Adverse Events (AEs) | To be evaluated after injection in vaccinees vs. placebo during the 7-day follow-up period of each injection (day of administration and 6 following days)
  Number of participants with solicited AEs, including local and general post-injection
Safety - Unsolicited AEs | To be evaluated after injection in vaccinees vs. placebo during the 28-day follow-up period after each injection (day of administration and 27 following days)
  Number of participants with unsolicited AEs post-injection
Safety - All Solicited and Unsolicited AEs post-injection | To be evaluated after injection in vaccinees vs. placebo during the 28-day follow-up period after each injection (day of administration and 27 following days)
  Number of participants with any AEs post-injection
Safety - Unsolicited AEs post-challenge | To be evaluated after challenge in vaccinees vs. placebo during the 28-day follow-up period post-challenge (day of challenge and 27 following days)
  Number of participants with unsolicited AEs post-challenge
Safety - Medically relevant AEs post-injection | To be evaluated in vaccinees vs. placebo from 28 days post each injection until receipt of next injection, challenge, or until their study end
  Number of participants with medically relevant AEs post-injection
Safety - Medically relevant AEs post-challenge | To be evaluated in vaccinees vs. placebo from 28 days post-challenge (Day 57) until their study end
  Number of participants with medically relevant AEs post-challenge
Safety - Serious Adverse Events (SAEs) | To be evaluated after injection in vaccinees vs. placebo until their study end
  Number of participants with SAEs
Safety - AEs leading to withdrawal from the trial | To be evaluated after injection in vaccinees vs. placebo until their study end
  Number of participants with AEs leading to withdrawal from the trial
Safety - Evaluate changes in hematological and blood chemistry parameters following injection | To be evaluated at 7-days of each post-injection compared to baseline values in vaccinees vs. placebo
  Number of participants with hematological and blood chemistry laboratory abnormalities
Immunogenicity - Geometric mean titers (GMTs) of anti-S. sonnei LPS IgGs in serum | To be evaluated in vaccinees vs. placebo from Day 1 until study end
  Anti-S. sonnei LPS IgG titer in serum collected at V1, V2, V3, V4, V5/a/b, V6, V7 and V8 in Step 1, and at V1, V2, V3, V4, C-1, C8, and V6 in Step 2
Immunogenicity - GMTs of anti-S. flexneri 2a LPS IgGs in serum | To be evaluated in vaccinees vs. placebo from Day 1 until study end
  Anti-S. flexneri 2a LPS IgG titer in serum collected at V1, V2, V3, V4, V5/a/b, V6, V7 and V8 in Step 1, and at V1, V2, V3, V4, C-1, C8, and V6 in Step 2
Immunogenicity - GMTs of anti-S. flexneri 3a LPS IgGs in serum | To be evaluated in vaccinees vs. placebo from Day 1 until study end
  Anti-S. flexneri 3a LPS IgG titer in serum collected at V1, V2, V3, V4, V5/a/b, V6, V7 and V8 in Step 1, and at V1, V2, V3, V4, C-1, C8, and V6 in Step 2
Immunogenicity - GMTs of anti-S. flexneri 6 LPS IgGs in serum | To be evaluated in vaccinees vs. placebo from Day 1 until study end
  Anti-S. flexneri 6 LPS IgG titer in serum collected at V1, V2, V3, V4, V5/a/b, V6, V7 and V8 in Step 1, and at V1, V2, V3, V4, C-1, C8, and V6 in Step 2
Immunogenicity - establish or confirm immunomarker that correlate with a reduced risk of shigellosis | To be evaluated in challenged vaccinees from Day 1 to Day 65
  Association between the primary shigellosis outcome and each of the following:
  * Serum anti-S. sonnei LPS IgG titer at C-1 (pre-challenge)
  * Maximum post-vaccination serum anti-S. sonnei LPS IgG titer through C-1 (pre-challenge)
  * Fold change from V1 (baseline) to C-1 (pre-challenge) in serum anti-S. sonnei LPS IgG titer
Immunogenicity - establish or confirm immunomarker that correlate with a reduced risk of moderate-to-severe shigellosis | To be evaluated in challenged vaccinees from Day 1 to Day 65
  Association between moderate-to-severe shigellosis and each of the following:
  * Serum anti-S. sonnei LPS IgG titer at C-1 (pre-challenge)
  * Maximum post-vaccination serum anti-S. sonnei LPS IgG titer through C-1 (pre-challenge)
  * Fold change from V1 (baseline) to C-1 (pre-challenge) in serum anti-S. sonnei LPS IgG titer
Immunogenicity - establish or confirm immunomarker that correlate with a reduced risk of solicited events | To be evaluated in challenged vaccinees from Day 1 to Day 65
  Association between the occurrence (any severity) and severity of each solicited event following challenge and each of the following:
  * Serum anti-S. sonnei LPS IgG titer at C-1 (pre-challenge)
  * Maximum post-vaccination serum anti-S. sonnei LPS IgG titer through C-1 (pre-challenge)
  * Fold change from V1 (baseline) to C-1 (pre-challenge) in serum anti-S. sonnei LPS IgG titer

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar R Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Paulina A Rebolledo, MD, Principal Investigator — Emory University; Robert W Frenck, Jr., MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Hope Clinic of Emory University, Atlanta, Georgia
  - Johns Hopkins Center for Immunization Research, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarkson KA, Talaat KR, Alaimo C, Martin P, Bourgeois AL, Dreyer A, Porter CK, Chakraborty S, Brubaker J, Elwood D, Frolich R, DeNearing B, Weerts HP, Feijoo B, Halpern J, Sack D, Riddle MS, Fonck VG, Kaminski RW. Immune response characterization in a human challenge study with a Shigella flexneri 2a bioconjugate vaccine. EBioMedicine. 2021 Apr;66:103308. doi: 10.1016/j.ebiom.2021.103308. Epub 2021 Apr 1. PMID 33813141
- [Background] Cohen D, Ashkenazi S, Green MS, Gdalevich M, Robin G, Slepon R, Yavzori M, Orr N, Block C, Ashkenazi I, Shemer J, Taylor DN, Hale TL, Sadoff JC, Pavliakova D, Schneerson R, Robbins JB. Double-blind vaccine-controlled randomised efficacy trial of an investigational Shigella sonnei conjugate vaccine in young adults. Lancet. 1997 Jan 18;349(9046):155-9. doi: 10.1016/S0140-6736(96)06255-1. PMID 9111538
- [Background] Cohen D, Ashkenazi S, Green M, Lerman Y, Slepon R, Robin G, Orr N, Taylor DN, Sadoff JC, Chu C, Shiloach J, Schneerson R, Robbins JB. Safety and immunogenicity of investigational Shigella conjugate vaccines in Israeli volunteers. Infect Immun. 1996 Oct;64(10):4074-7. doi: 10.1128/iai.64.10.4074-4077.1996. PMID 8926071
- [Background] Frenck RW Jr, Dickey M, Suvarnapunya AE, Chandrasekaran L, Kaminski RW, Clarkson KA, McNeal M, Lynen A, Parker S, Hoeper A, Mani S, Fix A, Maier N, Venkatesan MM, Porter CK. Establishment of a Controlled Human Infection Model with a Lyophilized Strain of Shigella sonnei 53G. mSphere. 2020 Sep 23;5(5):e00416-20. doi: 10.1128/mSphere.00416-20. PMID 32968005
- [Background] Hausdorff WP, Anderson JD 4th, Bagamian KH, Bourgeois AL, Mills M, Sawe F, Scheele S, Talaat K, Giersing BK. Vaccine value profile for Shigella. Vaccine. 2023 Nov 3;41 Suppl 2:S76-S94. doi: 10.1016/j.vaccine.2022.12.037. Epub 2023 Oct 10. PMID 37827969
- [Background] Kotloff KL, Riddle MS, Platts-Mills JA, Pavlinac P, Zaidi AKM. Shigellosis. Lancet. 2018 Feb 24;391(10122):801-812. doi: 10.1016/S0140-6736(17)33296-8. Epub 2017 Dec 16. PMID 29254859
- [Background] MacLennan CA, Aguilar AO, Steele AD. Consensus Report on Shigella Controlled Human Infection Model: Introduction and Overview. Clin Infect Dis. 2019 Dec 9;69(Suppl 8):S577-S579. doi: 10.1093/cid/ciz886. PMID 31816066
- [Background] MacLennan CA, Grow S, Ma LF, Steele AD. The Shigella Vaccines Pipeline. Vaccines (Basel). 2022 Aug 24;10(9):1376. doi: 10.3390/vaccines10091376. PMID 36146457
- [Background] Martin P, Alaimo C. The Ongoing Journey of a Shigella Bioconjugate Vaccine. Vaccines (Basel). 2022 Jan 29;10(2):212. doi: 10.3390/vaccines10020212. PMID 35214671
- [Background] Passwell JH, Ashkenazi S, Banet-Levi Y, Ramon-Saraf R, Farzam N, Lerner-Geva L, Even-Nir H, Yerushalmi B, Chu C, Shiloach J, Robbins JB, Schneerson R; Israeli Shigella Study Group. Age-related efficacy of Shigella O-specific polysaccharide conjugates in 1-4-year-old Israeli children. Vaccine. 2010 Mar 2;28(10):2231-2235. doi: 10.1016/j.vaccine.2009.12.050. Epub 2010 Jan 5. PMID 20056180
- [Background] Porter CK, Thura N, Ranallo RT, Riddle MS. The Shigella human challenge model. Epidemiol Infect. 2013 Feb;141(2):223-32. doi: 10.1017/S0950268812001677. Epub 2012 Aug 21. PMID 22906296
- [Background] Porter CK, Lynen A, Riddle MS, Talaat K, Sack D, Gutierrez RL, McKenzie R, DeNearing B, Feijoo B, Kaminski RW, Taylor DN, Kirkpatrick BD, Bourgeois AL. Clinical endpoints in the controlled human challenge model for Shigella: A call for standardization and the development of a disease severity score. PLoS One. 2018 Mar 28;13(3):e0194325. doi: 10.1371/journal.pone.0194325. eCollection 2018. PMID 29590182
- [Background] Riddle MS, Kaminski RW, Di Paolo C, Porter CK, Gutierrez RL, Clarkson KA, Weerts HE, Duplessis C, Castellano A, Alaimo C, Paolino K, Gormley R, Gambillara Fonck V. Safety and Immunogenicity of a Candidate Bioconjugate Vaccine against Shigella flexneri 2a Administered to Healthy Adults: a Single-Blind, Randomized Phase I Study. Clin Vaccine Immunol. 2016 Dec 5;23(12):908-917. doi: 10.1128/CVI.00224-16. Print 2016 Dec. PMID 27581434
- [Background] Talaat KR, Alaimo C, Martin P, Bourgeois AL, Dreyer AM, Kaminski RW, Porter CK, Chakraborty S, Clarkson KA, Brubaker J, Elwood D, Frolich R, DeNearing B, Weerts H, Feijoo BL, Halpern J, Sack D, Riddle MS, Fonck VG. Human challenge study with a Shigella bioconjugate vaccine: Analyses of clinical efficacy and correlate of protection. EBioMedicine. 2021 Apr;66:103310. doi: 10.1016/j.ebiom.2021.103310. Epub 2021 Apr 13. PMID 33862589